CLINICAL TRIAL: NCT03012451
Title: Measuring the Health and Wellbeing Impacts of a Scalable Program of Psychosocial Intervention for Refugee Youth
Brief Title: A Psychosocial Program Impact Evaluation in Jordan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Queen Margaret University (Other); University of Western Ontario, Canada (Other); Harvard University (Other); University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1502015359
Record Dates: First submitted 2016-12-21; First posted 2017-01-06 (Estimated); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Stress, Psychological; Mental Health Impairment
Keywords: Stress; Insecurity; Mental Health
MeSH Terms: conditions — Stress, Psychological; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Advancing Adolescents (Experimental): Received structured eight-week psychosocial sessions
  Interventions: Behavioral: Advancing Adolescents
- Control (No Intervention): Controls wait-listed for the intervention, matched for age and urban residence

INTERVENTIONS:
Behavioral: Advancing Adolescents — The "Advancing Adolescents" programme is a structured 8-week psychosocial intervention for adolescents in humanitarian crises, based on profound stress attunement processes. It features three elements that are widely viewed as important to support youth adjustment in contexts of complex emergencies: (i) safety: establishment of a 'safe space' within the community as a base for activities and site of protection; (ii) support: facilitation of social support and self-expression; and (iii) structured activities: access to scheduled group activities.
  Arms: Advancing Adolescents

SUMMARY:
The study aims to deliver a robust pre-post evaluation of the wellbeing impacts of an innovative, brief, and scalable psychosocial intervention, delivered to refugee youth living in urban settlements in Jordan. The study was conducted using two waves of data collection: the first featured an intervention and a matched control group, the second featured a full randomized control trial.

DETAILED DESCRIPTION:
This study will provide a robust evaluation of the Mercy Corps 'Advancing Adolescents, No Lost Generation' program that targets stress alleviation in refugee youth (12-18 years) with specific measures of psychosocial stress, biological stress, and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Eligible and enrolled in Mercy Corps Advancing Adolescents program
* Syrian refugee and Jordanian host-community youth residing in 4 urban centers in northern Jordan

Exclusion Criteria:

* Not available for study recruitment (started sessions or deferred sessions before study start date).

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 817 (Actual)
Dates: Start 2015-04; Primary Completion 2016-09 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Psychosocial Stress: Insecurity (Regional Measure) | 11 weeks
  Insecurity was measured with The Human Insecurity (HI). This tool was developed for use in the West Bank (Ziadni, Hammoudeh et al. 2011, Hamayel, Ghandour et al. 2014). The 10-item scale is a 5-point Likert scale with scores expressed as percentages on a scale of 0-100. The HI covers issues such as worries regarding inability to obtain daily life necessities, losing a source of income, fears about the future, and family safety.
Psychosocial stress: Distress (Regional Measure) | 11 weeks
  Distress was measured with the Human Distress scale (Hamayel & Ghandour, 2014), developed for use with conflict-affected adolescents in the West Bank. The 12-item scale is a 5-point Likert scale with scores expressed as percentages on a scale of 0-100. Sample items include, "To what extent have you felt worried," "To what extent did you feel humiliated," and "To what extent did you feel angry." Scores are presented as percentages (0-100%), with higher scores indicating greater distress.
Psychosocial Stress (International Measure) | 11 weeks
  Stress was measured using the Arabic version of the Perceived Stress Scale (Cohen, Karmarck, & Mermelstein, 1983), validated with a Jordanian sample (Almadi, Cathers, Hamdan Mansour, & Chow, 2012). This 14-item, 5-point Likert scale measures perceived stress over the last month, with higher scores indicating greater stress. Items include, "How often have you been upset because of something that happened unexpectedly?" and "How often have you been able to control irritations in your life?" (reverse-scored) (1 = Never, 5 = Very often).

SECONDARY OUTCOMES:
Mental Health Difficulties: Regional Measure | 11 weeks
  Mental health was assessed using the 21-item Arab Youth Mental Health questionnaire (Mahfoud et al., 2011; Mahkoul et al., 2011). This measure includes questions such as, "During the last week I was upset", "During the last week I was bored and hated my life", and "During the last week, I was having a lot of headaches, stomach-aches, and nausea" (1 = Rarely, 3 = Always). Higher scores indicate more symptoms of anxiety and depression.
Mental Health Difficulties: International Measure | 11 weeks
  The Arabic version of the Strengths and Difficulties Questionnaire (SDQ), a brief screening tool for psychiatric difficulties (Alyahri & Goodman, 2006) was used. The 20 items include emotional, conduct, and hyperactivity symptom scores (range 0-40). We summed score of the Arabic version of the SDQ subscales relating to hyperactivity, emotional symptoms, conduct problems, and peer problems (Alyahri & Goodman, 2006).
Prosocial Behavior: International Measure | 11 weeks
  The Strengths and Difficulties Questionnaire (SDQ) Prosocial Score, which featured 5 items to assess prosociality was used. Items include "I try to be nice to other people. I care about their feelings" and "I am helpful if someone is hurt, upset, or feeling sick" (0 = Not true, 2 = Certainly true). Higher scores indicate greater prosociality.
Resilience: Cross-cultural Measure | 11 weeks
  Resilience was measured using the CYRM-28 (Liebenberg et al., 2012; Ungar & Liebenberg, 2011), which had been translated and culturally grounded for use into Arabic. Responses ranged from 1 ("Not at all") to 5 ("A lot"), with higher scores indicating greater resilience.
Biological Stress: Cortisol | 11 weeks
  Cortisol was obtained from immunoassays of scalp hair cortisol that provide useful measures of the altered activity of the hypothalamic-pituitary-adrenal axis. Scalp hair is collected non-invasively (~100 strands, 0.5 cm area). This measure indicates chronic stress over the last month, and examined per individual for pre/post intervention levels. These analyses are being undertaken by Professor van Uum at Western Ontario University.
Biological Stress: Cell-mediated Immune Function | 11 weeks
  Cell-mediated immune function was measured in field settings, using systemic suppression of immune function in response to chronic stress is measured via immunoassays for Epstein Barr Virus antibodies, in conjunction with C-Reactive Protein, from dried blood spots collected from pricking the finger with a sterile disposable lancet. Three drops of blood on filter paper are dried at room temperature, then frozen until lab assay. This measure reflects compromised immune response due to psychosocial stress over the past week, and examined per individual for pre/post intervention levels.
Cognitive function | 11 weeks
  Cognitive function was assessed using tablet-based cognitive skill tasks, testing hippocampal function (long term memory) and prefrontal executive function. Children play short games (1-4 min each) during which they press the tablet in response to geometric shapes. Responses during game play are recorded and used to measure cognitive function.

OTHER OUTCOMES:
Posttraumatic stress symptoms | 11 weeks
  The Arabic version of the Child Revised Impact of Events Scale (CRIES-8, 4-point scale) was implemented to assess posttraumatic stress symptoms. Analysis will be on dimensional scores, noting that CRIES >17 points is predictive of symptoms of posttraumatic stress disorder (http://www.childrenandwar.org).
Genetic markers of trauma and/or stress | 11 weeks
  Genetic and epigenetic analyses in DNA will be undertaken from cheek swab samples to investigate the biological signatures of altered expressions of trauma and/or psychosocial stress. Whole-genome amplification of the extracted DNA will be used to generate maximum genetic data from the samples.

CONTACTS AND LOCATIONS:
Overall Officials: catherine panter-brick, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
We are sharing the anonymized dataset with project collaborators, but only with other researchers upon explicit request.

REFERENCES:
- [Derived] Panter-Brick C, Dajani R, Eggerman M, Hermosilla S, Sancilio A, Ager A. Insecurity, distress and mental health: experimental and randomized controlled trials of a psychosocial intervention for youth affected by the Syrian crisis. J Child Psychol Psychiatry. 2018 May;59(5):523-541. doi: 10.1111/jcpp.12832. Epub 2017 Oct 2. PMID 28967980
- See also: Save the Children Fund Enhancing Learning and Research for Humanitarian Assistance — http://www.elrha.org/map-location/yale-psychosocial-call2/